CLINICAL TRIAL: NCT05828316
Title: The Impact of a Resilience-based Intervention on Emotional Regulation, Grit and Life Satisfaction: A Comparative Study Between Egyptian and Saudi Nursing Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4112023
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2022-04

CONDITIONS: Resilience-based Intervention, Emotional Regulation, Grit and Life Satisfaction
MeSH Terms: conditions — Emotional Regulation; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 60 students (30 nursing students in alexandria- 30 nursing students in Saudi). They will participate in resilience based intervention
  Interventions: Behavioral: Resilience-based intervention
- Control group (No Intervention): 60 students (30 nursing students in alexandria- 30 nursing students in Saudi). They will not participate in resilience based intervention

INTERVENTIONS:
Behavioral: Resilience-based intervention — resilience-based intervention is a curriculum that offers a careful selection of evidence-based exercises to build coping skills and promote thriving. The resilience-based intervention philosophy is that there are many routes to achieving greater resiliency. Each participants choose from a menu of exercises in the areas of goal-setting, emotional skills, social connection, health, meaning, and self-talk. The ability to choose exercises that fit their specific goals, interests, and schedules is important, because the most effective strategies are the ones that people actually do, which tend to be the ones that are most enjoyable and personally relevant. No single practice is going to work for everyone regardless of its proven benefits. resilience-based intervention makes improving well-being accessible, manageable and fun, by introducing a variety of bite-sized, exercises that participants can experiment with and find what works for them.
  Arms: Intervention group

SUMMARY:
Nursing students may be perceived as having a stable college experience because they have a relatively clear career goal and a higher employment rate than students in other majors, but they consistently report that their heavy study loads, frequent exams, and clinical practice cause them to feel more stressed and depressed than students in other majors (Chernomas & Shapiro 2013, Lee & Jang 2021). Focusing on emotional events that have a direct impact on nursing students' learning and the college experience is crucial to their psychological wellbeing (Lee & Jang 2021). In order to improve the emotional experiences and life satisfaction of nursing students, it is crucial to determine the factors that affect their emotions.

DETAILED DESCRIPTION:
A constructivist and grounded theory design was recently used to create a model of resilience for nursing students (Reyes et al. 2015). Three steps represent how resilience is experienced, according to the "Pushing Through" model of resilience: first, "stepping into," or embracing, the adversity. The second is "staying the course," or understanding that they must keep working toward their objectives. Finally, "acknowledge" what they have learned from their difficulties and how they feel prepared to face new challenges. Additionally, students had brief obstacles, such as 'disengaging' from class because they felt overburdened. This paradigm serves as a lens to illustrate how, despite facing challenges, resilience can be developed over time. There is early support for encouraging resilience in nursing students before they begin their professions given the data linking resilience to burnout in nursing students

ELIGIBILITY:
Inclusion Criteria:

* nursing students who are willing to participate in the study and don't have any psychiatric illnesses

Exclusion Criteria:

* Those who refuse to participate in the study, nursing students with psychiatric illnesses

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-05 (Estimated)

PRIMARY OUTCOMES:
The Emotion Regulation Questionnaire (ERQ) | 2 weeks
  It is a 10-item self-report scale designed to assess the habitual use of two commonly used strategies to alter emotion: cognitive reappraisal and expressive suppression. Participants respond to each item using a 7-point Likert scale ranging from 1 n(strongly disagree) to 7 (strongly agree). Cognitive reappraisal involves thinking differently about a situation in order to change its meaning in order to alter one's emotional experience. Expressive suppression involves decreasing the outward expression of emotion. Six items contribute to the subscale for cognitive reappraisal (e.g., "When I'm faced with a stressful situation, I make myself think about it in a way that helps me stay calm"). Four items contribute to the subscale for expressive suppression (e.g., "When I am feeling negative emotions, I make sure not to express them") (Gross, & John 2003).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No